CLINICAL TRIAL: NCT06415695
Title: Evaluating the Feasibility of a Dietary Weight Loss Program to Overcome Obesity and Its Comorbidity Among Arab Populations: Pilot Study
Brief Title: Evaluating the Feasibility of a Dietary Weight Loss Program to Overcome Obesity and Its Comorbidity Among Arab Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asma Yahya (Other)
Collaborators: King Abdullah Medical City (Other Government)
Responsible Party: Sponsor-Investigator, Asma Yahya, Doctoral Student - Main Investigator, University of Illinois at Urbana-Champaign
Organization: University of Illinois at Urbana-Champaign (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB23-0344
Record Dates: First submitted 2024-04-23; First posted 2024-05-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
Keywords: Online weight loss program; Feasibility assessment; Dietary education; Sustainable weight loss; Pilot study
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The interventional study model for this research involves implementing a single-group, pre-post design to assess the effectiveness of a three-month weight loss intervention among participants with a body mass index (BMI) over 25 kg/m². Participants will engage in ten weekly online sessions covering topics related to dietary and lifestyle improvements. The intervention will be delivered through educational materials specifically tailored for the Saudi population and accessed via an online platform. Participants will also receive a Wi-Fi-enabled scale for self-monitoring of their weight loss progress throughout the intervention period. Data collection will include surveys, dietary assessments, physical measurements, and lifestyle habit assessments at baseline and three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-group, pre-post design to evaluate a three-month weight loss intervention in adult. (Experimental): Ten 40-minute education sessions appropriate to Saudi people will be developed and will cover essential topics for enhancing diet, lifestyle, and health. Each session comprises four modules, including activities and homework reviewed by a dietitian. Based on the EMPOWER weight loss program developed by the Nakamura lab for the US population, adjustments will be made to align with Saudi preferences, including food choices and cooking methods. Participants will access these materials online.
  Interventions: Behavioral: Education sessions

INTERVENTIONS:
Behavioral: Education sessions — Ten 40-minute education sessions appropriate to Saudi people will be developed and will cover essential topics for enhancing diet, lifestyle, and health. Each session comprises four modules, including activities and homework reviewed by a dietitian. Based on the EMPOWER weight loss program developed by the Nakamura lab for the US population, adjustments will be made to align with Saudi preferences, including food choices and cooking methods. Participants will access these materials online.

SUMMARY:
This study aims to develop and test a culturally tailored online weight loss program for the Saudi population. Building upon the success of a previous program in the United States, the research team will adapt educational materials and conduct a pilot study to assess the feasibility and initial outcomes of the program among Arab participants. The study seeks to answer questions about the program's acceptability, effectiveness, and scalability, with the ultimate goal of combating obesity and its related health issues in Saudi Arabia.

DETAILED DESCRIPTION:
This research project aims to help Saudi individuals lose weight in a way that suits their culture. Obesity is a significant problem and can lead to serious health issues like diabetes and heart problems. Even though Saudi Arabia has attempted to help individuals lose weight before, previous efforts haven't been successful enough. Therefore, the investigators aim to develop a new weight loss program that is better suited to Saudi individuals.

First, educational materials will be created in Arabic to teach individuals how to eat better and live healthier. Then, collaboration will be undertaken with individuals in Saudi Arabia to ensure the program fits their needs. Afterward, the program will be tested with a small group of individuals to evaluate its effectiveness and acceptability.

Approximately 20 individuals will be invited to join the program at King Abdullah Medical City. They will participate in ten online sessions, where they will learn about healthy eating and lifestyle improvements. Additionally, they will regularly weigh themselves. Data will be collected before and after the program to assess its impact on weight loss and overall well-being.

By the end of the project, the investigators hope to have developed an effective program that assists Saudi individuals in losing weight and maintaining good health.

ELIGIBILITY:
Inclusion Criteria:

* Adults within the age range of 18 to 75 years old
* Individuals with a BMI greater than 25 kg/m²
* Proficient in the Arabic language
* Not currently pregnant or breastfeeding
* Not using glucagon-like peptide -1 (GLP-1) or any weight loss medications
* Have not undergone bariatric surgery
* Possess Wi-Fi connectivity at their residence
* Own a smartphone
* Willing to provide consent for participation in 10 educational sessions spanning three months.

Exclusion Criteria:

* Individuals not meeting the inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-23 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Program feasibility and acceptability | 3 months
  Participants' views on the program's feasibility and acceptability will be gauged through structured surveys or interviews at the intervention's end.
  We'll employ two surveys:
  Feasibility Survey: this survey developed based on a previous study, examines various aspects like personal gain, program content, and engagement. Participants rate questions on a 1-5 scale and provide open-ended feedback.
  Feedback Survey: Participants will rate enjoyment, likelihood of recommendation, perceived benefits, and willingness to pay for services on a 1-5 scale. Open-ended questions will capture additional feedback.

SECONDARY OUTCOMES:
Weight Loss | 3 months
  Change in body weight from baseline to three months.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah Medical City (KAMC), Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
IPD won't be shared due to privacy and confidentiality concerns.